CLINICAL TRIAL: NCT02431221
Title: A Study on the Efficacy, Safety, and Tolerability of Perhexiline Maleate in Subjects With Hypertrophic Cardiomyopathy and Moderate-To-Severe Heart Failure
Brief Title: Efficacy, Safety, and Tolerability of Perhexiline in Subjects With Hypertrophic Cardiomyopathy and Heart Failure
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of efficacy in a preceding study.
Sponsor: Heart Metabolics Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HM-PHX-003
Record Dates: First submitted 2015-04-27; First posted 2015-04-30 (Estimated); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Hypertrophic Cardiomyopathy
Keywords: perhexiline; HCM; Hypertrophic Cardiomyopathy; CPEX
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — Perhexiline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Perhexiline maleate will be supplied in 100 mg and 25 mg tablets. It will be initially administered at a dose of 200 mg once a day in tablet form for at least six months. After initiation of dosing, perhexiline dosing will be determined using plasma level guided dose adjustment. Dosing decisions will be made by an unblinded dose control center.
  Interventions: Drug: Perhexiline
- Placebo (Placebo Comparator): Placebo will be administered once a day in tablet form for at least six months. Tablets will be identical in size and shape to perhexiline tablets. Adjustments in placebo dosing will be made by an unblinded dose control center to mimic decisions made for subjects in the experimental arm.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Perhexiline — perhexiline maleate, oral, 25mg or 100mg tablets Whenever initiating PHM therapy, subjects will receive a loading regimen of PHM as indicated in in the Heart Metabolics Dose Justification document. Drug levels will be measured first on Day 4 +/- 1 day, with an initial dose adjustment performed on Day 7 +/- 1 day, as needed. The next sampling will occur on Day 21 +/- 1 day for potential dose adjustment, as advised by the DCC, on or about Day 24. Subsequent dosing will be monitored and advised by a Dose Control Center
  Arms: Intervention
Drug: Placebo
  Arms: Placebo

SUMMARY:
A Study on the Efficacy, Safety, and Tolerability of Perhexiline maleate in Subjects with Hypertrophic Cardiomyopathy and Moderate-To-Severe Heart Failure

DETAILED DESCRIPTION:
This study is an international, multi-center, randomized, double-blind, placebo controlled clinical trial of the effects of perhexiline maleate on a rank-ordered, hierarchical variable consisting of outcome and functional measures in 350 subjects with hypertrophic cardiomyopathy and symptoms of moderate to severe congestive heart failure. The study is designed in four parts: 1) an open-label run-in period of 2 weeks, 2) A blinded, randomized phase of variable duration (anticipated between 6 months and 18 months depending on enrollment rate), 3) an open label period of 3 months, and 4) a randomized withdrawal period of 3 months. Subjects who do not experience an adverse outcome (death or resuscitated ventricular arrhythmia, stroke, need for surgical intervention, cardiovascular hospitalization, occurrence of atrial fibrillation, or study dropout) will undergo cardiopulmonary exercise testing in order to determine change from baseline in maximum oxygen consumption.

ELIGIBILITY:
Inclusion Criteria:

General Criteria

1. Adult, at least 18 years of age
2. Able and willing to give written informed consent Cardiomyopathy-related Criteria
3. Hypertrophic cardiomyopathy (HCM) with moderate-to-severe heart failure as defined as meeting all of the following criteria:

   1. HCM meeting the 2011 ACCF/AHA Criteria for the Diagnosis of Hypertrophic Cardiomyopathy (Gersh et al. 2011)
   2. Left ventricular hypertrophy (LVH) with maximum LV wall thickness > 15 mm by echocardiography or cardiac magnetic resonance imaging without an alternative explanation
   3. Left ventricular ejection fraction (LVEF) > 40%
   4. Able to perform exercise testing but unable to exceed 75% of the predicted age-adjusted maximum level(as determined by METs achieved during exercise testing-eligibility is not based on VO2max)
4. Normal sinus rhythm at Screening and Baseline (atrial fibrillation pattern acceptable for subjects with known chronic atrial fibrillation)
5. If taking any medications for the treatment of HCM (including beta-blockers, calcium channel blockers, disopyramide, diuretics), the medication has been taken a stable dose for at least 60 days prior to enrollment and will be continued at the same dose throughout the study

Exclusion Criteria:

General Criteria

1. Pregnant women, women who intend to become pregnant, or woman who are not practicing contraception, either pharmacologically or with a barrier method
2. Lactating women
3. CYP2D6 Poor Metabolizer (PM) status, based on genotype known prior to Screening, or as predicted by genotype assessed at Screening CYP2D6 Poor Metabolizer (PM) status is defined as having no functional CYP2D6 alleles by genotyping (exclusively having allele combinations of *3, *4, *5, *6, *7, *8, *12, *14).
4. Any subject who regularly takes a medication known to be a strong inhibitor of CYP2D6 (bupropion, fluoxetine, paroxetine, quinidine, or ritonavir)
5. Any concomitant disease, condition, or treatment that could interfere with the conduct of the study, or that would, in the opinion of the investigator or sponsor, pose an unacceptable risk to subjects and/or interfere with the interpretation of study data, including but not limited to:

   1. History of a known toxic or inflammatory peripheral neuropathy, such as mononeuritis multiplex, acute or chronic inflammatory demyelinating polyneuropathy (AIDP or CIDP), axonal sensorimotor neuropathies, drug-related neuropathy or neuritis, or diabetic neuropathy (history of a compression neuropathy, such as carpal tunnel syndrome, is acceptable)
   2. Poorly controlled diabetes mellitus (e.g., HbA1c > 8.5%)
   3. Clinically severe chronic obstructive pulmonary disease (i.e. COPD requiring home oxygen or history of IV or oral steroid use)
   4. History of a known chronic liver disease including cirrhosis of any cause, or chronic hepatitis B or hepatitis C
   5. History of porphyria
   6. History of recurrent hypoglycemia
   7. Active infection requiring antibiotics
   8. Life expectancy of less than 2 years
   9. Evidence of an active or suspected cancer or a history of malignancy, except for skin squamous cell or basal cell carcinomas that did not require systemic therapy and are considered to be cured
   10. History of substance abuse, including alcohol or illicit drugs within the past 12 months
   11. Abnormal safety studies of clinical significance at Screening such as:

   i. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase, or lactate dehydrogenase > 1.5X upper limit of normal (ULN)

   ii. Glucose < 70 mg/dL iii. Prolonged QTc (>450 msec) l. Known hypersensitivity to perhexiline maleate
6. Unable or unwilling to comply with the protocol
7. Enrolled in another therapeutic trial for hypertrophic cardiomyopathy

   Cardiomyopathy-related Exclusion Criteria
8. Asymptomatic subjects or subjects whose symptoms are controlled with medications
9. Resting LVOT gradient > 50 mmHg or known exercise-induced LVOT gradient > 80 mmHg
10. Absence of an implanted, operational ICD if there is a history of frequent non-sustained ventricular tachycardia, or a first degree relative having had sudden cardiac death or ICD implant
11. Known coronary artery disease (> 50% arterial luminal narrowing of a major epicardial vessel)
12. History of cardiac transplantation
13. Cardiac surgery or septal reduction surgery planned or having occurred within past 6 months
14. HCM believed to be caused by infiltrative disorders, glycogen storage disorders, and hypertensive heart disease (including genotypic or phenotypic evidence of Fabry's Disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Subject Outcome Variable | 6 months after randomization
  The subject Outcome variable is a rank-ordered, hierarchical classification of outcome variables followed by a rank ordering of change from baseline in Maximum oxygen consumption

SECONDARY OUTCOMES:
Functional Assessment During Randomized Withdrawal Phase | 6 months after initiation of open label period, and 3 months after randomized withdrawal period initiated
  Change of CPEX-VO2max from the beginning of the Randomized Withdrawal phase to the end of the Randomized Withdrawal phase (Part 4). The change in CPEX-VO2max in the placebo group will be compared to the change in CPEX-VO2max in the continued perhexiline (non-withdrawal) group.
Functional Assessment During Randomized Phase | 6 months after Randomization
  Change in six-minute walk test (6MWT) from baseline (pre-Part 1 run-in, prior to receiving any perhexiline) to 6 months after randomization during the Randomized Treatment (Part 2)
Functional Assessment During Randomized Withdrawal Phase | 6 months after initiation of open label period, and 3 months after randomized withdrawal period initiated
  Change in six-minute walk test (6MWT) from the beginning of the Randomized Withdrawal (Part 4) to the end of the Randomized Withdrawal (Part 4)